CLINICAL TRIAL: NCT06888726
Title: Efficacy of High-Intensity Transcranial Alternating Current Stimulation (Hi-tACS) in Treating Negative Symptoms of Schizophrenia
Brief Title: Efficacy of Hi-tACS for Schizophrenia Negative Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-TX-021
Record Dates: First submitted 2025-02-20; First posted 2025-03-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia; Negative Type; Transcranial Alternating Current Stimulation
Keywords: Hi-tACS; Schizophrenia; Randomized Controlled Trial; Negative symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: In this study, the RAND function in Excel is used to generate a random number table to form the random group assignment sequence, which is simple randomization. Interventions are standardized by medical personnel who have passed a training test. Stimulation devices of two groups are identical in appearance. Blinding: The assessors, medical personnel and participants are blinded; the research coordinator assigned the enrolled schizophrenia patients to the Hi-tACS intervention group or the sham stimulation control group based on the randomization table. The assessors, medical personnel and participants are not informed of the treatment group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- intervention group (Experimental): On the basis of maintaining regular medication, the intervention group received continuous Hi-tACS stimulation. The intervention was administered twice daily, in the morning and afternoon, from Monday to Friday for 2 weeks, with each session lasting 40 minutes, totaling 20 sessions.
  Interventions: Device: High-intensity transcranial alternating current stimulation (Hi-tACS)
- control group (Sham Comparator): On the basis of maintaining regular medication, the control group received sham Hi-tACS stimulation, with each stimulation session lasting only 40 seconds. The intervention was administered twice daily, in the morning and afternoon, from Monday to Friday for 2 weeks, with each session lasting 40 minutes, totaling 20 sessions.
  Interventions: Device: Sham High-intensity transcranial alternating current stimulation (Sham-Hi-tACS)

INTERVENTIONS:
Device: High-intensity transcranial alternating current stimulation (Hi-tACS) — The equipment used is the transcranial microcurrent stimulator (Nexalin ADI), operated by trained therapists following standardized instructions. Three Nexalin conductive electrodes are placed on the patient's head. A 4.45×9.53 cm electrode is placed on the forehead, corresponding to the Fpz region of the 10/20 international standard electrode placement system. Two 3.18×3.81 cm electrodes are placed on the bilateral dorsolateral prefrontal cortex, corresponding to the F3 and F4 regions of the international standard electrode placement system. The stimulation frequency is 77.5 Hz, and the current intensity is 15 mA.
  Arms: intervention group
Device: Sham High-intensity transcranial alternating current stimulation (Sham-Hi-tACS) — A sham device looks exactly the same as Nexalin ADI is used.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to investigate whether Hi-tACS is effective and safe in treating negative symptoms of schizophrenia.

Schizophrenic patients will receive treatment (Hi-tACS or shame stimulation) for 2 weeks.

Negative symptoms, cognitive functioning, social functioning, and quality of life of intervention group and control group were assessed and compared between the two groups at baseline, 2 weeks, and 3 months post-intervention.

DETAILED DESCRIPTION:
Objective: To investigate the therapeutic effects and short-term and long-term efficacy of high-intensity transcranial alternating current stimulation (Hi-tACS) on negative symptoms of schizophrenia.

Methods: A randomized controlled design was used, 60 schizophrenic patients who met the enrollment criteria were randomly assigned to either the Hi-tACS intervention group or the sham stimulation control group. Both groups continued their regular medication regimen. The intervention group received continuous current stimulation, while the control group received only 40 seconds of current stimulation per session. The treatment was administered twice daily (morning and afternoon) from Monday to Friday for 2 weeks, with each session lasting 40 minutes, for a total of 20 sessions. Negative symptoms, cognitive function, social function, and quality of life were assessed at baseline, 2 weeks, and 3 months post-intervention.

The primary outcome will be clinical symptoms, the secondary outcome will be the social function and quality of life, and the process measures included social cognition and neurocognition.

ELIGIBILITY:
Inclusion Criteria:

* Han Chinese population;
* Age ≥ 18 years;
* Education level ≥ 6 years, able to fill out questionnaires on their own, and having sufficient audiovisual level to complete the necessary examinations;
* Meets DSM-5 diagnostic criteria for schizophrenia as assessed by MINI 7.0;
* Residual negative symptoms, with at least one item ≥2 on the negative subscale of PANSS (N1-N7);
* Taking second-generation atypical antipsychotic medication, with no medication or dosage adjustments in the last two weeks
* Patients and guardians agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Meets DSM-5 diagnostic criteria for other mental disorders;
* Total score ≥19 on the PANSS positive subscales (P1-P7) ;
* Severe negative symptoms that prevent the patient from completing the required assessments and interventions;
* Serious physical or central nervous system disease (intracranial infection, intracranial tumor, presence of metal objects in the skull; epilepsy, seizures; history of hydrocephalus or central nervous system tumors; with implanted electronic devices; serious cardiac disease and fitted with a pacemaker, etc.);
* Impaired skin integrity at the site of electrode placement or hypersensitivity to electrode gels or adhesives;
* Mental retardation (Wechsler Adult Intelligence Scale WAIS <70) and/or severe cognitive impairment (Brief Mental State Examination MMSE <24);
* Presence of vision and/or hearing problems that prevent completion of relevant tests;
* Alcohol or drug abuse/dependence;
* Pregnancy;
* Those who have participated or are participating in other clinical studies 3 months ago;
* Failure or refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in negative symptoms of schizophrenia | change between baseline (W0), the end of intervention at 2 weeks (W2) and 3 months after intervention (M3)
  The primary efficacy evaluation measure is the Positive and Negative Syndrome Scale (PANSS), with statistical parameters including the PANSS total score and the negative subscale score. These scores reflect the severity of schizophrenia symptoms, with higher total or subscale scores indicate more severe symptoms. A decrease in scores after the intervention indicates symptom reduction and effective intervention.

SECONDARY OUTCOMES:
Change in sleep quality of clinical symptom | change between baseline (W0), the end of intervention at 2 weeks (W2) and 3 months after intervention (M3)
  The sleep quality assessment measure is Pittsburgh Sleep Quality Index (PSQI). The PSQI is a widely used self-report questionnaire designed to assess sleep quality over a one-month period. The PSQI consists of 19 items, which are grouped into seven components. Each component is scored on a scale from 0 to 3, with higher scores indicating worse sleep quality. The total score ranges from 0 to 21, and a higher total score suggests poorer overall sleep quality. A decrease in the total score after the intervention suggests an improvement in sleep quality.
Change in depression of clinical symptom | change between baseline (W0), the end of intervention at 2 weeks (W2) and 3 months after intervention (M3)
  The depression assessment measure is Hamilton Depression Rating Scale (HAMD). The HAMD is a widely used tool for assessing the severity of depression in individuals. The HAMD consists of 17 items. Each item is rated on a scale ranging from 0 to 4 or 0 to 2, with higher scores indicating more severe symptoms. A decrease in the total score after the intervention suggests an improvement in depression.
Change in anxiety of clinical symptom | change between baseline (W0), the end of intervention at 2 weeks (W2) and 3 months after intervention (M3)
  The anxiety assessment measure is Hamilton Anxiety Scale (HAMA). The HAMA is a 14-item scale designed to assess the severity of anxiety symptoms in individuals. The total score ranges from 0 to 56, with higher scores indicating greater anxiety severity. A decrease in the total score after the intervention suggests an improvement in anxiety.
Change in theory of mind of social cognition | change from baseline (W0) to 3 months after intervention (M3)
  The theory of mind assessment measure is faux pas recognition (FPT). The FPT examines the patient's recognition of the faux pas situation of the speaker. Higher total scores on the FTP indicate a better ability to recognize and understand faux pas, as well as stronger empathetic skills. An increase in the total score after the intervention suggests an improvement in theory of mind and social cognition.
Change in emotion perception of social cognition | change from baseline (W0) to 3 months after intervention (M3)
  The emotion perception assessment measure is Face Emotion Identification Task (FEIT). The FEIT assesses the ability to perceive emotions. The score ranges from 0 to 30, with higher scores indicating better emotion perception. An increase in the total score after the intervention suggests an improvement in emotion perception.
Change in coping styles of social cognition | change from baseline (W0) to 3 months after intervention (M3)
  The coping styles assessment measure is Simplified Coping Style Questionnaire (SCSQ). The SCSQ assesses the coping styles of individuals when facing setbacks. The overall coping style score is typically calculated as the difference between the positive coping score and the negative coping score. A higher overall score suggests a more proactive and positive coping style. An increase in the total score after the intervention suggests an improvement in positive coping style.
Change in attributional styles of social cognition | change from baseline (W0) to 3 months after intervention (M3)
  The attributional styles assessment measure is Attributional Style Questionnaire (ASQ). The ASQ assesses attributional styles. Each cause of 12 events was rated according to locus of control (internal vs. external), stability, and globality, with higher scores indicating greater attractiveness on each dimension and a score of 4 indicating a neutral response. An increase in internal, stable, and global dimensions for positive events and a decrease in these dimensions for negative events after the intervention suggests an improvement in attributional styles.
Change in neuropsychological status of cognitive function | change between baseline (W0), the end of intervention at 2 weeks (W2) and 3 months after intervention (M3)
  The neuropsychological status of cognitive function assessment measure is the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). The RBANS is widely used in clinical settings to detect cognitive impairments and track cognitive changes over time. It consists of 12 subtests that assess five primary cognitive domains: immediate memory, visuospatial/constructional skills, attention, language and delayed memory. The total RBANS score is derived by summing the five index scores and then converting this sum to a total scale score using the provided normative tables. The total scale score ranges from 40 to 160, with higher scores indicating better cognitive function. An increase in the total score after the intervention suggests an improvement in neuropsychological status of cognitive function.
Change in EEG data of cognitive function | change between baseline (W0), the end of intervention at 2 weeks (W2) and 3 months after intervention (M3)
  The electroencephalogram (EEG) data of cognitive function is P300. The P300 has been widely used in research and clinical settings to assess cognitive function. It is characterized by a positive deflection in the EEG signal that typically occurs approximately 300 milliseconds after the presentation of a target stimulus. The P300 is typically elicited using an oddball paradigm, where infrequent target stimuli are interspersed among more frequent non-target stimuli. To measure the P300, EEG data are collected using a set of electrodes placed on the scalp according to the international 10-20 system. The data are then pre-processed to remove artifacts and segmented into epochs around the stimulus onset. The average ERP is calculated for target and non-target stimuli separately, and the P300 is identified within the 250-500 ms time window.
Change in social function | change from baseline (W0) to 3 months after intervention (M3)
  The social function assessment measure is the Personal and Social Performance scale (PSP). The PSP is a widely used observer-rated scale for assessing patients' social functioning. The scale primarily assesses four areas of functioning in patients: useful activities in society, personal and social relationships, self-care and disruptive and aggressive behaviors. After scoring each of the four areas separately, a total score is determined according to the scoring standards. The total score ranges from 0 to 100 points and is divided into 10 levels, with higher scores reflecting better social function and interpersonal relationships. An increase in post-intervention scores indicates an improvement in social function.
Change in quality of life | change from baseline (W0) to 3 months after intervention (M3)
  The quality of life assessment measure is the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). The SF-36 scale is used to assess patients' health-related quality of life. It comprises 8 subscales with a total of 36 items, covering both physical and mental health aspects. The raw scores of each subscale are converted into standard scores ranging from 0 to 100, with higher scores indicating better quality of life in that particular domain. An increase in post-intervention scores suggests an improvement in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No